CLINICAL TRIAL: NCT07401342
Title: An Assessment of the Efficacy and Safety of Employing a Duosomal Chemical Peel for Aesthetic Enhancement in the Periocular and Facial Regions
Acronym: AESEDCPAEPFR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2023/11/02
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chemical Peeling
Keywords: Chemoexfoliation; Skin Resurfacing; Topical Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants aged over 21 years included in the study (Experimental): They will receive an application of salicylic acid to the facial surface through continuous massaging for a duration of five minutes, facilitating the exfoliation of the superficial epidermal layers. Subsequently, a specific medication will be administered based on the skin characteristics and the intended treatment objective: salicylic acid for individuals predisposed to oily skin and acne, mandelic acid for those with irregular pigmentation and hyperpigmentation, lactic acid for individuals with sensitive skin, and glycolic acid for those with wrinkles and pigmentation changes due to aging. A moisturizer will then be applied and massaged continuously, allowing it to act for five minutes. These treatments will be administered weekly over a four-week period
  Interventions: Drug: Duosomal chemical peel application

INTERVENTIONS:
Drug: Duosomal chemical peel application — They will receive an application of salicylic acid to the facial surface through continuous massaging for a duration of five minutes, facilitating the exfoliation of the superficial epidermal layers. Subsequently, a specific medication will be administered based on the skin characteristics and the intended treatment objective: salicylic acid for individuals predisposed to oily skin and acne, mandelic acid for those with irregular pigmentation and hyperpigmentation, lactic acid for individuals with sensitive skin, and glycolic acid for those with wrinkles and pigmentation changes due to aging. A moisturizer will then be applied and massaged continuously, allowing it to act for five minutes. These treatments will be administered weekly over a four-week period.

SUMMARY:
This study will employ an experimental, prospective, longitudinal, and comparative before-and-after design. The objective is to assess the efficacy and safety of duosomal chemical peels as agents for enhancing the aesthetic appearance of the periocular and facial regions

DETAILED DESCRIPTION:
Participants aged over 21 years will be included in the study. They will receive an application of salicylic acid to the facial surface through continuous massaging for a duration of five minutes, facilitating the exfoliation of the superficial epidermal layers. Subsequently, a specific medication will be administered based on the skin characteristics and the intended treatment objective: salicylic acid for individuals predisposed to oily skin and acne, mandelic acid for those with irregular pigmentation and hyperpigmentation, lactic acid for individuals with sensitive skin, and glycolic acid for those with wrinkles and pigmentation changes due to aging. A moisturizer will then be applied and massaged continuously, allowing it to act for five minutes. These treatments will be administered weekly over a four-week period. Improvement as reported by the study participants will be evaluated using the Face-Q and SASSQ (Scientific Assessment Scale of Skin Quality) questionnaires. The SASSQ is an objective scale completed by the researcher, assessing loss of elasticity, wrinkles, roughness, pigmentation, erythema, and pore size on a scale from 0 to 4, where 0 denotes absence of the parameter and 4 indicates very severe changes. The FACE-Q is a subjective scale completed by the participants, ranging from 1 to 4, where 1 signifies very dissatisfied and 4 signifies very satisfied. Descriptive statistics of the demographic variables will be conducted, and analytical statistics using the Wilcoxon test will be employed to compare baseline and final results at the conclusion of the treatment. A p-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 21 years and older, both male and female, who seek enhancement of the periocular and facial regions will be considered for recruitment. Participants must agree to the study conditions, consent to the follow-up period as proposed, and provide informed consent for the procedure.

Exclusion Criteria:

* Individuals with psychiatric disorders, those exhibiting symptoms indicative of body dysmorphia, and those who have undergone facial filler treatments within the six months preceding the procedure. Elimination criteria: Participants who fail to adhere to follow-up protocols during the designated periods; those who receive additional treatments such as mesotherapy, botulinum toxin, chemical peeling, or facial fillers in the same area during the follow-up period; and those who, during the follow-up period, develop any debilitating illness or conditions resulting in a wasting/emaciation syndrome.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Objective skin quality improvement | From enrollment to the end of treatment at 4 weeks
  The SASSQ (Scientific Assessment Scale of Skin Quality) is an objective scale completed by the researcher, assessing loss of elasticity, wrinkles, roughness, pigmentation, erythema, and pore size on a scale from 0 to 4, where 0 denotes absence of the parameter and 4 indicates very severe changes
Subjective skin quality improvement | From enrollment to the end of treatment at 4 weeks
  The FACE-Q is a subjective scale completed by the participants, ranging from 1 to 4, where 1 signifies very dissatisfied and 4 signifies very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmologia F.A.P. Conde de Valenciana, I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From May to July 2026

REFERENCES:
- [Result] Garg VK, Sinha S, Sarkar R. Glycolic acid peels versus salicylic-mandelic acid peels in active acne vulgaris and post-acne scarring and hyperpigmentation: a comparative study. Dermatol Surg. 2009 Jan;35(1):59-65. doi: 10.1111/j.1524-4725.2008.34383.x. Epub 2008 Dec 8. PMID 19076192
- [Result] Gunn J, Holt CM, Francis SE, Shepherd L, Grohmann M, Newman CM, Crossman DC, Cumberland DC. The effect of oligonucleotides to c-myb on vascular smooth muscle cell proliferation and neointima formation after porcine coronary angioplasty. Circ Res. 1997 Apr;80(4):520-31. doi: 10.1161/01.res.80.4.520. PMID 9118483
- [Result] Lasic DD, Papahadjopoulos D. Liposomes revisited. Science. 1995 Mar 3;267(5202):1275-6. doi: 10.1126/science.7871422. No abstract available.
- [Result] Maher D. Tuberculosis is important problem in children with HIV infection in sub-Saharan Africa. BMJ. 1996 Aug 31;313(7056):562-3. doi: 10.1136/bmj.313.7056.562d. No abstract available. PMID 8790012
- [Result] Sarkar R, Garg V, Bansal S, Sethi S, Gupta C. Comparative Evaluation of Efficacy and Tolerability of Glycolic Acid, Salicylic Mandelic Acid, and Phytic Acid Combination Peels in Melasma. Dermatol Surg. 2016 Mar;42(3):384-91. doi: 10.1097/DSS.0000000000000642. PMID 26859648
- [Result] Odrzywolek W, Deda A, Zdrada J, Wilczynski S, Blonska-Fajfrowska B, Lipka-Trawinska A. Quantitative Evaluation of the Effectiveness of Chemical Peelings in Reducing Acne Lesions Based on Gray-Level Co-Occurrence Matrix (GLCM). Clin Cosmet Investig Dermatol. 2022 Sep 12;15:1873-1882. doi: 10.2147/CCID.S375131. eCollection 2022. PMID 36117771
- [Result] Grimes PE. The safety and efficacy of salicylic acid chemical peels in darker racial-ethnic groups. Dermatol Surg. 1999 Jan;25(1):18-22. doi: 10.1046/j.1524-4725.1999.08145.x. PMID 9935087
- [Result] Sharquie KE, Al-Tikreety MM, Al-Mashhadani SA. Lactic acid chemical peels as a new therapeutic modality in melasma in comparison to Jessner's solution chemical peels. Dermatol Surg. 2006 Dec;32(12):1429-36. doi: 10.1111/j.1524-4725.2006.32352.x. PMID 17199649
- [Result] Jarzabek-Perz S, Mucha P, Rotsztejn H. Corneometric evaluation of skin moisture after application of 10% and 30% gluconolactone. Skin Res Technol. 2021 Sep;27(5):925-930. doi: 10.1111/srt.13044. Epub 2021 Mar 26. PMID 33769633
- [Result] Dayal S, Kalra KD, Sahu P. Comparative study of efficacy and safety of 45% mandelic acid versus 30% salicylic acid peels in mild-to-moderate acne vulgaris. J Cosmet Dermatol. 2020 Feb;19(2):393-399. doi: 10.1111/jocd.13168. Epub 2019 Sep 25. PMID 31553119
- [Result] Yamamoto K, Oishi K, Fujimatsu I, Komatsu K. Production of R-(-)-mandelic acid from mandelonitrile by Alcaligenes faecalis ATCC 8750. Appl Environ Microbiol. 1991 Oct;57(10):3028-32. doi: 10.1128/aem.57.10.3028-3032.1991. PMID 1660699
- [Result] O'Connor AA, Lowe PM, Shumack S, Lim AC. Chemical peels: A review of current practice. Australas J Dermatol. 2018 Aug;59(3):171-181. doi: 10.1111/ajd.12715. Epub 2017 Oct 24. PMID 29064096
- [Result] Bensimon RH. Chemical Peels. Facial Plast Surg Clin North Am. 2023 Nov;31(4):475-494. doi: 10.1016/j.fsc.2023.05.006. Epub 2023 Jul 26. PMID 37806681
- [Result] Salam A, Dadzie OE, Galadari H. Chemical peeling in ethnic skin: an update. Br J Dermatol. 2013 Oct;169 Suppl 3:82-90. doi: 10.1111/bjd.12535. PMID 24098904
- [Result] Gentili G, Perugini P, Bugliaro S, D'Antonio C. Efficacy and safety of a new peeling formulated with a pool of PHAs for the treatment of all skin types, even sensitive. J Cosmet Dermatol. 2023 Feb;22(2):517-528. doi: 10.1111/jocd.15215. Epub 2022 Aug 9. PMID 35796684
- [Result] Roberts WE. Chemical peeling in ethnic/dark skin. Dermatol Ther. 2004;17(2):196-205. doi: 10.1111/j.1396-0296.2004.04020.x. PMID 15113287
- [Result] Asilian A, Shahmoradi Z, Talakoub M, Mokhtari F, Siadat AH, Mohaghegh F, Adibi N, Mozafarpoor S, Kazemipour S, Danesh F, Hafezi H. Evaluation of combination therapy with peeling added to minimal invasive blepharoplasty in lower eyelid rejuvenation. J Cosmet Dermatol. 2020 Nov;19(11):2922-2928. doi: 10.1111/jocd.13394. Epub 2020 Apr 3. PMID 32243049
- [Result] Dayan SH, Bacos JT, Ho TT, Gandhi ND, Gutierrez-Borst S, Kalbag A. Topical skin therapies in subjects undergoing full facial rejuvenation. J Cosmet Dermatol. 2019 Jun;18(3):798-805. doi: 10.1111/jocd.12977. Epub 2019 Apr 29. PMID 31033162
- [Result] Eiben-Nielson C, Kerscher M. Development and validation of a global photonumeric scale for evaluating skin quality of aged female facial skin. J Cosmet Dermatol. 2021 Dec;20(12):4032-4039. doi: 10.1111/jocd.14058. Epub 2021 Mar 24. PMID 33690945
- [Result] Kang MC, Lee JW, Lee TH, Subedi L, Wahedi HM, Do SG, Shin E, Moon EY, Kim SY. UP256 Inhibits Hyperpigmentation by Tyrosinase Expression/Dendrite Formation via Rho-Dependent Signaling and by Primary Cilium Formation in Melanocytes. Int J Mol Sci. 2020 Jul 28;21(15):5341. doi: 10.3390/ijms21155341. PMID 32731326
- [Result] Murase D, Hachiya A, Amano Y, Ohuchi A, Kitahara T, Takema Y. The essential role of p53 in hyperpigmentation of the skin via regulation of paracrine melanogenic cytokine receptor signaling. J Biol Chem. 2009 Feb 13;284(7):4343-53. doi: 10.1074/jbc.M805570200. Epub 2008 Dec 18. PMID 19098008
- [Result] Gao L, Song W, Qian L, Zhang J, Li K, Yang J, Wang G. Clinical efficacy of different therapeutic modes of CO2 fractional laser for treatment of static periocular wrinkles in Asian skin. J Cosmet Dermatol. 2022 Mar;21(3):1045-1050. doi: 10.1111/jocd.14640. Epub 2021 Dec 8. PMID 34889041